CLINICAL TRIAL: NCT03225846
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 1b/2a Study of WVE-120102 Administered Intrathecally in Patients With Huntington's Disease
Brief Title: Safety and Tolerability of WVE-120102 in Patients With Huntington's Disease
Acronym: PRECISION-HD2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: WVE-HDSNP2-001
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-01

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- WVE-120102 (2 mg) or placebo (Experimental)
  Interventions: Drug: WVE-120102; Drug: Placebo
- WVE-120102 (4 mg) or placebo (Experimental)
  Interventions: Drug: WVE-120102; Drug: Placebo
- WVE-120102 (8 mg) or placebo (Experimental)
  Interventions: Drug: WVE-120102; Drug: Placebo
- WVE-120102 (16 mg) or placebo (Experimental)
  Interventions: Drug: WVE-120102; Drug: Placebo
- WVE-120102 (32 mg ) or placebo (Experimental)
  Interventions: Drug: WVE-120102; Drug: Placebo

INTERVENTIONS:
Drug: WVE-120102 — WVE-120102 is a stereopure antisense oligonucleotide (ASO)
Drug: Placebo — 0.9% Sodium Chloride

SUMMARY:
PRECISION-HD2 is a Phase 1b/2a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple doses of WVE-120102 in adult patients with early manifest Huntington's disease (HD) who carry a targeted single nucleotide polymorphism (SNP) rs362331 (SNP2).

ELIGIBILITY:
Key Inclusion Criteria:

* Prescreened with targeted SNP on the same allele as the pathogenic CAG expansion
* Ambulatory, male or female patients aged ≥25 - ≤65 years
* Clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score = 4
* Early manifest HD, Stage I or Stage II based on UHDRS Total Functional Capacity Scores ≥7 and ≤13

Key Exclusion Criteria:

* Malignancy or received treatment for malignancy, other than treated basal cell or squamous cell carcinoma of the skin, within the previous 5 years
* Received investigational drug or implantable device in prior 3 months or investigational oligonucleotide in prior 6 months or 5 halflives of the oligonucleotide, whichever is longer
* Clinically significant medical condition, unstable psychiatric symptoms, substance abuse, or pregnancy
* Inability to undergo brain MRI
* Bone, spine, bleeding, or other disorder that exposes the patient to risk of injury or unsuccessful lumbar puncture

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (26):
- United States (5):
  - University of California San Diego, La Jolla, California
  - University of California Davis Medical Center, Sacramento, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (7):
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Melbourne Hospital, Carlton, Victoria
  - Monash Health, Clayton, Victoria
  - Alfred Health, Melbourne, Victoria
  - Calvary Health Care Bethlehem, Parkdale, Victoria
  - North Metropolitan Health Service, Perth, Western Australia
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Centre For Movement Disorders, Toronto, Ontario
  - Centre Hospitalier de l-Universite de Montreal, Montreal, Quebec
- Denmark (3):
  - Aarhus Universitets Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense University Hospital and University of Southern Denmark, Odense
- France (2):
  - Hospital Henri Mondor, Créteil
  - Institut du Cerveau et de la Moelle Epinière, Paris
- George-Huntington-Institut GmbH, Münster, Germany
- Poland (2):
  - Szpital Sw. Wojciecha, Gdansk
  - Instytut Psychiatrii i Neurologii, Warsaw
- United Kingdom (3):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Queen Elizabeth University Hospital - PPDS, Glasgow, Glasgow City
  - Royal Liverpool University Hospital, Liverpool

REFERENCES:
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: April 2020. J Huntingtons Dis. 2020;9(2):185-197. doi: 10.3233/JHD-200002. PMID 32250312
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: February 2018. J Huntingtons Dis. 2018;7(1):89-98. doi: 10.3233/JHD-189001. PMID 29480210

RESULTS

PARTICIPANT FLOW:
Groups:
- Pooled Placebo: Placebo: 0.9% Sodium Chloride
- WVE-120102 (2 mg); WVE-120102 (4 mg); WVE-120102 (8 mg); WVE-120102 (12 mg); WVE-120102 (16 mg); WVE-120102 (32 mg ): WVE-120102: WVE-120102 is a stereopure antisense oligonucleotide (ASO)
Period: Overall Study
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Started | 22 | 9 | 12 | 15 | 8 | 9 | 13
Single Dose Period Only | 6 | 3 | 4 | 7 | 8 | 0 | 4
Multiple Dose Period Only | 3 | 0 | 3 | 6 | 0 | 0 | 4
Single Dose and Multiple Dose | 13 | 6 | 5 | 2 | 0 | 9 | 5
Completed | 22 | 7 | 11 | 15 | 8 | 9 | 6
Not Completed | 0 | 2 | 1 | 0 | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Patient did not wish to comply with IC/EC | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Patient decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg ) | Total
Number analyzed (Participants) | 22 | 9 | 12 | 15 | 8 | 9 | 13 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (10.16) | 52.4 (11.59) | 46 (10.63) | 49.3 (10.40) | 47.1 (8.48) | 53.1 (8.33) | 54.1 (8.88) | 50.3 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 7 | 10 | 4 | 2 | 6 | 42
  Male | 14 | 4 | 5 | 5 | 4 | 7 | 7 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 21 | 9 | 12 | 15 | 8 | 9 | 13 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 22 | 9 | 12 | 15 | 8 | 9 | 13 | 88
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 8 | 2 | 1 | 0 | 6 | 0 | 26
  Denmark | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 5
  Poland | 4 | 0 | 4 | 3 | 0 | 1 | 1 | 13
  United Kingdom | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 4
  Australia | 2 | 0 | 0 | 0 | 0 | 0 | 7 | 9
  France | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Germany | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 5
  United States | 6 | 1 | 3 | 7 | 8 | 0 | 0 | 25
Time since initial diagnosis [Mean (Standard Deviation); unit: Years] | 6.1 (5.95) | 9.9 (8.80) | 3.8 (3.62) | 5.6 (2.80) | 3.9 (3.23) | 3.2 (5.61) | 5.6 (9.28) | 5.3 (6.21)
Age at disease onset [Mean (Standard Deviation); unit: Years] | 40.18 (10.527) | 42.00 (16.363) | 41.75 (12.129) | 43.33 (9.378) | 42.50 (9.289) | 49.00 (6.652) | 48.08 (12.796) | 44.47 (11.410)
Diagnosis stage [Count of Participants; unit: Participants] — Stage of disease, as defined by United Huntington's Disease Rating Scale, Total Functional Capacity Score. Stage 1 (least severe) = scores of 11 to 13. Stage 2 = scores of 7 to 10. Stages go up to Stage 5 = score of 0.
  Participants
    Stage 1 | 9 | 5 | 6 | 8 | 1 | 5 | 11 | 45
    Stage 2 | 13 | 4 | 6 | 7 | 7 | 4 | 2 | 43

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Patients With Treatment-emergent Adverse Events (TEAEs)
Description: All TEAEs reported or observed during the study, including TEAEs resulting from concurrent illnesses, reactions to concurrent medications, or progression of disease states
Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Population: No statistical analysis has been performed on these safety results
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 22 | 9 | 12 | 15 | 8 | 9 | 13
Participants | 20 | 8 | 9 | 13 | 4 | 8 | 13

2. Primary Outcome: Safety: Number of Patients Who Experienced Severe TEAEs
Description: Number of patients who experienced a severe treatment-emergent adverse event. Severity was evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Population: No statistical analysis has been performed on these safety results
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 22 | 9 | 12 | 15 | 8 | 9 | 13
Participants | 2 | 1 | 1 | 2 | 0 | 2 | 9

3. Primary Outcome: Safety: Number of Patients With Serious TEAEs
Description: A serious TEAE is defined as any event that results in death, is immediately life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect not present at Prescreening.
Time Frame: Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Population: No statistical analysis has been performed on these safety results
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 22 | 9 | 12 | 13 | 4 | 8 | 13
Participants | 0 | 1 | 2 | 2 | 0 | 0 | 9

4. Primary Outcome: Safety and Tolerability: Number of Patients Who Withdraw Due to TEAEs
Time Frame: Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Population: No statistical analysis has been performed on these safety results
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 22 | 9 | 12 | 15 | 8 | 9 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 6

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax)
Description: Cmax of WVE-120102 in plasma
Time Frame: Patients participating in Period 1 (SAD) had PK samples collected on Day 1 predose through 24-48 hours postdose. Patients participating in Period 2 (MAD) had PK samples collected predose on Day 112 and through 4 hours postdose.
Population: Overall number of participants analyzed represents patients with at least 1 postdose plasma or CSF measurement at Day 1. The overall number for Day 112 was different and represents patients with at least 1 postdose plasma or CSF measurement at Day 112. Specimen samples collected following administration of 12 mg dose were not analyzed or tested, and therefore no data are available to be reported for this Arm/Group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 9 | 9 | 9 | 0 | 9 | 9
ng/mL
  Day 1 | 1.35 (2.714) | 8.54 (6.073) | 29.87 (31.891) |  | 31.49 (15.801) | 96.21 (57.394)
  Day 112: number analyzed (Participants) | 6 | 8 | 8 | 0 | 9 | 0
  Day 112 | 7.46 (15.411) | 15.55 (14.587) | 36.16 (30.012) |  | 59.49 (35.718) |

6. Secondary Outcome: PK: Time of Occurrence of Cmax (Tmax)
Description: tmax of WVE-120102 in plasma
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Groups:
- WVE-120102 (12 mg): WVE-12101: WVE-120102 is a stereopure antisense oligonucleotide (ASO)
Arm/Group | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 9 | 9 | 9 | 0 | 9 | 9
hour
  Day 1 | 3.33 (7.742) | 1.26 (1.044) | 1.77 (1.101) |  | 1.77 (1.345) | 3.09 (3.752)
  Day 112: number analyzed (Participants) | 6 | 8 | 8 | 0 | 9 | 0
  Day 112 | 1.22 (0.314) | 1.86 (0.874) | 2.06 (1.206) |  | 1.98 (0.828) |

7. Secondary Outcome: PK: Area Under the Plasma Concentration-time Curve (AUC 0-t)
Description: AUC 0-t from time zero to the last quantifiable concentration of WVE-120102 in plasma
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 9 | 9 | 9 | 0 | 9 | 9
hr*ng/mL
  Day 1 | 24.65 (9.108) | 62.05 (67.358) | 132.44 (91.913) |  | 804.92 (1456.786) | 919.14 (271.997)
  Day 112: number analyzed (Participants) | 6 | 8 | 8 | 0 | 9 | 0
  Day 112 | 23.83 (23.187) | 35.47 (22.280) | 107.83 (70.198) |  | 133.22 (67.683) |

8. Secondary Outcome: PK: Terminal Elimination Half-life
Description: Terminal elimination half life of WVE-120102 in plasma (t1/2)
Time Frame: as for outcome 5
Population: The t1/2 value was calculated using data from patients who had at least 3 postdose concentration values in the terminal phase. No patients had sufficient postdose samples at Day 112 to calculate t1/2 values. Specimen samples collected following administration of 12 mg dose were not analyzed or tested, and therefore no data are available to be reported for this Arm/Group.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 0 | 2 | 1 | 0 | 5 | 6
hour |  | 33.42 (30.983) | 6.23 (NA) — Standard deviation is not applicable with an n=1 |  | 13.45 (4.604) | 18.17 (20.969)

9. Secondary Outcome: Pharmacodynamics (PD): Percentage Change From Baseline in Mutant Huntingtin Protein
Description: Percentage change from baseline to last observation in mutant huntingtin protein
Time Frame: Day 1 to last observation - up to Day 140 (32 mg cohort) or Day 196 (all other cohorts)
Population: The 12 mg dose group was not included in this analysis as these patients only received a single dose and did not attend the Day 140/Day 196 visit.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 16 | 6 | 8 | 8 | 9 | 8
Percent change from baseline | -2.64 [-14.89 to 11.71] | 3.46 [-7.67 to 7.80] | -3.53 [-4.20 to 2.41] | -3.45 [-6.46 to 7.35] | -5.82 [-12.09 to 6.44] | -2.06 [-28.72 to 7.84]

10. Secondary Outcome: Clinical Effects: Total Functional Capacity (TFC)
Description: Percentage change from baseline to the last measured time point in the Total Functional Capacity score, administered as part of the Unified Huntington's Disease Rating Scale (UHDRS). Total Functional Capacity is scored 13 (normal) to 0 (severe disability)
Time Frame: Day 1 Day 1 to last observation - up to Day 140 (32 mg cohort) or Day 196 (all other cohorts)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
Number analyzed (Participants) | 16 | 6 | 8 | 8 | 9 | 9
Percent change from baseline | 0.0 [0.00 to 0.00] | 0.0 [-2.00 to 0.00] | 0.0 [0.00 to 0.00] | -4.17 [-13.89 to 0.00] | -8.33 [-16.67 to 0.00] | 0.00 [0.00 to 0.00]

ADVERSE EVENTS:
Time Frame: Day 1 to end of study (Day 196 [32 mg cohort] or Day 210 [all other cohorts])
Arm/Group | Pooled Placebo | WVE-120102 (2 mg) | WVE-120102 (4 mg) | WVE-120102 (8 mg) | WVE-120102 (12 mg) | WVE-120102 (16 mg) | WVE-120102 (32 mg )
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/9 | 0/12 | 1/15 | 0/8 | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/9 | 2/12 | 2/15 | 0/8 | 0/9 | 9/13
Other Adverse Events (participants affected / at risk) | 22/22 | 9/9 | 12/12 | 15/15 | 8/8 | 9/9 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=22) | WVE-120102 (2 mg) (N=9) | WVE-120102 (4 mg) (N=12) | WVE-120102 (8 mg) (N=15) | WVE-120102 (12 mg) (N=8) | WVE-120102 (16 mg) (N=9) | WVE-120102 (32 mg ) (N=13)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=22) | WVE-120102 (2 mg) (N=9) | WVE-120102 (4 mg) (N=12) | WVE-120102 (8 mg) (N=15) | WVE-120102 (12 mg) (N=8) | WVE-120102 (16 mg) (N=9) | WVE-120102 (32 mg ) (N=13)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4 | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 3 | 2 | 3 | 1 | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 5 | 0 | 2 | 1 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 2 | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 5 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chemical burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
CSF protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Blood fibrinogen increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chest X-ray abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Complement factor C3 decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Complement factor C3 increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cells urine (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 5 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Athralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headace (Nervous system disorders) | 8 | 3 | 3 | 3 | 0 | 6 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 0 | 0 | 3 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cerebellar ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0 | 2 | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Loss of proprioception (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chorea (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Reflexes abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Abnormal behavior (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anger (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalized anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chronic throat clearing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03225846/Prot_SAP_000.pdf